CLINICAL TRIAL: NCT06788977
Title: CEFALY Pregnancy Registry
Brief Title: External Trigeminal Nerve Stimulation for Migraine Treatment in Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Cefaly Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: 51001
Record Dates: First submitted 2024-11-27; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy; Migraine; Headache; Postpartum; Depression; Anxiety
Keywords: Pregnancy; Migraine; Headache; Neuromodulation; Trigeminal Nerve Stimulation; External Trigeminal Nerve Stimulation; Postpartum; drug-free; medications; complementary therapy; alternative therapy; wholistic therapy; natural; non-invasive device
MeSH Terms: conditions — Migraine Disorders; Headache; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- External Trigeminal Nerve Stimulation (eTNS) group: This group reflects participants who are already using eTNS therapy during the pregnancy, as well as participants who start using eTNS therapy at any point during their pregnancy.
  Any participant may opt to continue or discontinue eTNS treatments during the registry period, which will not affect their ability to participate.
  Interventions: Device: external Trigeminal Nerve Stimulation
- Non-eTNS group: This group reflects participants who have not used eTNS therapy during and throughout their pregnancy. If a participant who initially does not use eTNS therapy during pregnancy decides to start eTNS therapy at any point during their pregnancy, they will be assigned to the eTNS group.

INTERVENTIONS:
Device: external Trigeminal Nerve Stimulation — External trigeminal nerve stimulation (e-TNS) is a non-invasive, nondrug option for the acute and preventative treatment of migraine. The device is marketed under the trade name CEFALY and has received clearance from the US Food and Drug Administration (FDA) for the acute and preventative treatment of migraine.
  The CEFALY device provides transcutaneous stimulation of the supraorbital and supratrochlear branches of the ophthalmic division of the Trigeminal nerve. Patients apply a self-adhesive electrode pad to their forehead, then place the CEFALY generator over the electrodes, resulting in a magnetic connection. The user then selects a treatment program for acute or preventative therapy, which lasts for 60 or 20 minutes.
  Other Names: supraorbital transcutaneous stimulator (STS)
  Groups: External Trigeminal Nerve Stimulation (eTNS) group

SUMMARY:
This online registry aims to understand the potential benefits and safety of external trigeminal nerve stimulation for the treatment of migraine in pregnant women. Women do not need to use external trigeminal nerve stimulation or any other form of migraine treatment to participate in the registry.

The main question it aims to answer is:

Is external trigeminal nerve stimulation a safe and effective option for migraine treatment during and after pregnancy?

There are no required changes in migraine treatment to participate in this registry. Participants may or may not use external trigeminal nerve stimulation or any other treatment they currently use and may still participate in the registry. There are no clinic or research visits, as the registry is entirely online. Participants will be asked to complete up to six 15- 20-minute surveys over a time period of up to 12 months.

DETAILED DESCRIPTION:
This will be a prospective research registry from which retrospective research studies will derive. Individuals who are eligible to participate in the CEFALY Pregnancy Registry will be pregnant women who have migraines or headaches. Use of the external Trigeminal Neurostimulation (eTNS) device is not mandatory for participation in the registry, and the registry will include information from individuals who use and do not use eTNS (CEFALY) to treat their migraines or headaches before, during, and after pregnancy.

The ideal candidate for participation will be women within 14 weeks gestation at the time of screening enrollment, as this will minimize any recall bias. However, women in the second and third trimesters during screening and enrollment will not be excluded and may also participate in the registry. The registry will aim to enroll 550 participants per the inclusion and exclusion criteria.

Registry participation, including consent, screening, enrollment, and completion of registry surveys, will be completed online using a confidential survey platform accessed via a publicly available web-based link. Once the simple consent is acknowledged, the potential participant will enter their name, email, phone number and date of birth. The phone number, and email entered are required to conduct the registry data collection process.

Participants will then complete screening questions to assess their eligibility for the registry. If they meet all eligibility requirements, they will be required to upload sufficient evidence of a current intrauterine pregnancy. The registry investigators will verify the uploaded document for accuracy before enrollment. The participant's name and date of birth are required to validate a current pregnancy based on the required uploaded documents during the screening process.

If eligible and documentation of current pregnancy is confirmed, the investigators will enroll the participant in the registry and start the survey process. Enrolled participants who have agreed to participate in the registry will receive an invitation to the requested surveys via automated email and short message service (SMS) text. The links provided in the email and SMS text will automatically direct the participant to the appropriate survey based on the timing of their enrollment, estimated due date, pregnancy status, and date of completion of prior surveys. Before each survey attempt, enrolled participants will need to verify their identity with an automated authentication code provided to their registered email address and phone number they provided during initial screening to verify their data and protect their entered health information.

In general, the surveys will ask questions about the participant's health history, their previous pregnancies (if applicable), current pregnancy, migraine or headache symptoms and migraine treatments and therapies. In addition, participants will be asked to complete several validated scales assessing the degree of migraine disability and mental health impact. If the participant indicates that they are using eTNS CEFALY during the registry process, they will also receive surveys about their eTNS use. Any unclear survey responses are found during periodic reviews as part of data quality assurance. In that case, study staff may contact the participant via email and/or phone call to clarify an answer or answers on the survey.

In most circumstances, the registry participants will be asked to complete up to six surveys. Based on preliminary registry testing, the enrollment (consent and screening) and baseline period will take participants approximately 20 minutes to complete. The five sets of surveys (1st, 2nd, 3rd trimester, early postpartum, and late postpartum) will take approximately 10 - 15 minutes for each participant to complete. Therefore, we estimate that the total participation time for most participants will be between 60 and 90 minutes. In some situations, the timing and number of surveys and time points requested will differ for some participants based on their responses.

A link to a survey will be sent to the participant's email and phone via text for each of the following time points as indicated by the patient's estimated due date at time of enrollment.

Pre-pregnancy and Baseline: This survey will be sent following registry enrollment First trimester: This survey will be sent at 14 weeks gestation Second trimester: This survey will be sent at 28 weeks gestation Third trimester: This survey will be sent at 37 weeks gestation. Early postpartum: This survey will be sent 6 weeks following childbirth Late postpartum: This survey will be sent 12 weeks following childbirth

If the participant enrolls in the registry beyond any of the gestation periods described above, they will also be asked to complete the baseline and earlier trimester surveys before their current trimester following registry enrollment. If the participant delivers before 37 weeks gestation, the third-trimester survey will be sent following notification of childbirth.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing and able to provide simple consent for registry participation.
2. Has access to email, text messages via smartphone or computer with internet access
3. Be between the ages of 18 to 44 years at enrollment.
4. Pregnant with one fetus/baby at time of enrollment (singleton pregnancy)
5. Have headaches or migraines prior to pregnancy and continued to have headaches or migraines into pregnancy OR headaches or migraines began while pregnant in the first trimester.
6. Able to provide proof of active intrauterine pregnancy and estimated due date, via online document upload, using any of the following documents:

   1. ultrasound report of current pregnancy
   2. beta hcg lab report
   3. a signed provider's medical documentation confirming intrauterine pregnancy with fetal heart sounds and estimated due date
   4. a signed provider's note on a prescription sheet or physician letterhead confirming intrauterine pregnancy and estimated due date

Exclusion Criteria:

1. Patients under the age of 18 or over the age of 44 at enrollment
2. Not pregnant at time of enrollment
3. Pregnant with more than one fetus/baby at time of enrollment (multigestational pregnancy)
4. Patients with any other condition which might preclude participation in the opinion of the patient's physician(s) or the study's principal investigator
5. No access to email, smartphone, or computer with internet access

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All participants in the registry should be (1) age 18-44 years, (2) pregnant with one fetus/baby at the time of enrollment (3) experience migraines or headaches during pregnancy or at the time of enrollment and (4) have access to email and text messages to receive notifications and reminders for registry surveys.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2030-11-27 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Rate of miscarriage per trimester | through study completion average 2 years
Postpartum Bonding according to the Maternal-to-Infant Bonding Scale | through study completion average 2 years
  The "Maternal-to-Infant Bonding Scale" is a scale which measures the mother's feelings regarding her child within the first few weeks after birth. The score of teh scale can range from 0 which denotes favorable or good outcome whereas the maximum score is 24 indicating a poor outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Deena Kuruvilla, MD, Principal Investigator
Locations (1):
- https://public.smart-trial.co/#/public/649d77f0e8f8d0fb993d0c61/6626f6a04f0a3c7dd0860e14/662726d84f0a3c7dd08aeaa0/signup?lang=en-us&enforceLanguage=true, Darien, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Given the potentially sensitive nature of the information collected within the registry, IPD will not be shared to protect participants' information as much as possible.

REFERENCES:
- [Background] Nappi RE, Tiranini L, Sacco S, De Matteis E, De Icco R, Tassorelli C. Role of Estrogens in Menstrual Migraine. Cells. 2022 Apr 15;11(8):1355. doi: 10.3390/cells11081355. PMID 35456034
- [Background] Skajaa N, Szepligeti SK, Xue F, Sorensen HT, Ehrenstein V, Eisele O, Adelborg K. Pregnancy, Birth, Neonatal, and Postnatal Neurological Outcomes After Pregnancy With Migraine. Headache. 2019 Jun;59(6):869-879. doi: 10.1111/head.13536. Epub 2019 May 8. PMID 31069791
- [Background] Frederick IO, Qiu C, Enquobahrie DA, Aurora SK, Peterlin BL, Gelaye B, Williams MA. Lifetime prevalence and correlates of migraine among women in a pacific northwest pregnancy cohort study. Headache. 2014 Apr;54(4):675-85. doi: 10.1111/head.12206. Epub 2013 Aug 28. PMID 23992560
- [Background] Welander NZ, Mwinyi J, Asif S, Schioth HB, Skalkidou A, Fransson E. Migraine as a risk factor for mixed symptoms of peripartum depression and anxiety in late pregnancy: A prospective cohort study. J Affect Disord. 2021 Dec 1;295:733-739. doi: 10.1016/j.jad.2021.08.119. Epub 2021 Sep 4. PMID 34517247
- [Background] Friedman LE, Aponte C, Perez Hernandez R, Velez JC, Gelaye B, Sanchez SE, Williams MA, Peterlin BL. Migraine and the risk of post-traumatic stress disorder among a cohort of pregnant women. J Headache Pain. 2017 Dec;18(1):67. doi: 10.1186/s10194-017-0775-5. Epub 2017 Jul 6. PMID 28685258
- [Background] Kuruvilla DE, Mann JI, Tepper SJ, Starling AJ, Panza G, Johnson MAL. Phase 3 randomized, double-blind, sham-controlled Trial of e-TNS for the Acute treatment of Migraine (TEAM). Sci Rep. 2022 Mar 24;12(1):5110. doi: 10.1038/s41598-022-09071-6. PMID 35332216
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Plummer F, Manea L, Trepel D, McMillan D. Screening for anxiety disorders with the GAD-7 and GAD-2: a systematic review and diagnostic metaanalysis. Gen Hosp Psychiatry. 2016 Mar-Apr;39:24-31. doi: 10.1016/j.genhosppsych.2015.11.005. Epub 2015 Nov 18. PMID 26719105
- [Background] Wood ME, Burch RC, Hernandez-Diaz S. Polypharmacy and comorbidities during pregnancy in a cohort of women with migraine. Cephalalgia. 2021 Mar;41(3):392-403. doi: 10.1177/0333102420975394. Epub 2020 Dec 3. PMID 33269942
- [Background] Burch R. Epidemiology and Treatment of Menstrual Migraine and Migraine During Pregnancy and Lactation: A Narrative Review. Headache. 2020 Jan;60(1):200-216. doi: 10.1111/head.13665. Epub 2019 Oct 3. PMID 31579938
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- See also: Headaches.com — https://www.headaches.com/